CLINICAL TRIAL: NCT02100527
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled Study To Evaluate The Safety, Tolerability And Effects Of PF-05175157 On Moderate To Severe Acne Vulgaris In Adult Subjects
Brief Title: Study Of Safety, Tolerability And Effects Of PF-05175157 In Adults With Moderate To Severe Acne Vulgaris
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study canceled
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1731019
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Acne Vulgaris
Keywords: safety; tolerability; pharmacokinetics; oral dosing; moderate to severe acne vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05175157 (Experimental)
  Interventions: Drug: PF-05175157
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — 200 mg (as 2x100 mg tablets) twice a day (BID) for 6 weeks
  Arms: PF-05175157
Drug: Placebo — placebo matching 200 mg (as 2x100 mg tablets) BID for 6 weeks
  Arms: Placebo

SUMMARY:
This is a 6 week study to characterize the safety, tolerability and effects of PF-05175157 administered for 6 weeks in subjects with moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years or older diagnosed with moderate to severe acne vulgaris who are otherwise healthy.
* Normal spirometry at screening (FEV1 and FVC (Forced Vital Capacity)at least 80% predicted).
* Minimum of 20 inflammatory lesions on the face.
* Willing to discontinue other acne treatments prior to and during the study period through follow-up.

Exclusion Criteria:

* Subjects with active nodulocystic acne.
* Subjects unwilling to comply with lifestyle guidelines, commit to study visits, and perform study procedures.
* History of dry eye or other known disease that affects the sclera or cornea.
* History of pulmonary disease or inability to adequately perform testing.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Weeks 2, 4, and 6
  Physical examination, pulmonary function testing, adverse event monitoring, ECGs, vital signs, laboratory tests

SECONDARY OUTCOMES:
Sebum measurements | Weeks 2, 4, and 6
  Change from baseline in amount and rate of sebum excretion
Pharmacokinetics of PF-05175157 | Weeks 2, 4, and 6
  Plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731019&StudyName=Study%20Of%20Safety%2C%20Tolerability%20And%20Effects%20Of%20PF-05175157%20In%20Adults%20With%20Moderate%20To%20Severe%20Acne%20Vulgaris